CLINICAL TRIAL: NCT07039123
Title: Polygenic Risk Score to Optimize Primary Prevention in Intermediate Risk Population (PERSONAL)
Brief Title: Polygenic Risk Score for Optimizing Primary Prevention in Intermediate-Risk Populations
Acronym: PERSONAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PERSONAL-2025-00601
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Primary Prevention of Cardiovascular Disease
Keywords: Polygenic risk score; Cardiovascular risk; Genomic medicine; Cardiovascular disease; Intermediate cardiovascular risk; Primary prevention; Genetic risk stratification
MeSH Terms: conditions — Genetic Risk Score; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Study nurse/Research Fellow providing the information of cardiovascular risk at baseline will be masked. Patients will be masked as both groups will receive genetic results (intervention group during the study, control group at the end of the study).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polygenic Risk Score Combined with SCORE2 (Experimental): Participants in this arm will receive cardiovascular risk assessment using a combination of traditional clinical risk factors (SCORE2 algorithm) and a polygenic risk score for coronary artery disease (PRS-CAD). The combined risk (PRS-CAD-SCORE2) will be communicated using a structured communication tool developed by the study team. Participants and their healthcare providers will receive the results, and those with elevated risk will be referred to a lipid consultation. Lifestyle guidance and educational materials will also be provided.
  Interventions: Diagnostic Test: Polygenic Risk Score for Coronary Artery Disease (PRS-CAD); Behavioral: Standardized Risk Communication Tool (SCORE2)
- SCORE2-Based Risk Assessment (Active Comparator): Participants in this arm will receive standard cardiovascular risk assessment using the SCORE2 algorithm only. Risk results will be communicated using the same structured communication tool, without inclusion of genetic information. No polygenic risk score will be calculated or disclosed. Participants and their healthcare providers will receive the standard risk results and general lifestyle recommendations.
  Interventions: Behavioral: Standardized Risk Communication Tool (SCORE2)

INTERVENTIONS:
Diagnostic Test: Polygenic Risk Score for Coronary Artery Disease (PRS-CAD) — A polygenic risk score will be calculated based on genome-wide genotyping and combined with SCORE2 clinical risk factors to estimate personalized cardiovascular risk. The combined risk (PRS-CAD-SCORE2) will be communicated to participants and their healthcare providers using a standardized communication tool. Participants with elevated risk will be referred to a lipid clinic.
  Arms: Polygenic Risk Score Combined with SCORE2
Behavioral: Standardized Risk Communication Tool (SCORE2) — Participants will receive risk communication based solely on clinical risk factors using the SCORE2 algorithm. The same structured communication tool will be used (without genetic data), along with general lifestyle guidance.

SUMMARY:
The goal of this clinical trial is to determine whether incorporating a polygenic risk score (PRS) can optimize primary cardiovascular disease prevention in individuals with intermediate cardiovascular risk.

The main questions it aims to answer are:

* Can a polygenic risk score improve risk stratification in intermediate-risk individuals?
* Does disclosing polygenic risk information to patients and physicians lead to better preventive interventions (e.g., statin use, lifestyle changes)? Researchers will compare outcomes in participants with PRS disclosure versus standard risk assessment to see if PRS-guided prevention leads to improved cardiovascular risk management.

Participants will:

* Undergo baseline cardiovascular risk assessment
* Provide a blood sample for PRS calculation
* Complete follow-up visits for lifestyle counseling, medication review, and risk reassessment

DETAILED DESCRIPTION:
Coronary artery disease (CAD) remains the leading cause of mortality worldwide. While current cardiovascular disease (CVD) prevention guidelines rely on clinical risk scores such as SCORE2, these tools may underestimate or overestimate risk in individuals with intermediate clinical risk. Polygenic risk scores (PRS) aggregate the effect of multiple common genetic variants and may provide additional predictive value when combined with traditional risk assessment.

This randomized controlled trial evaluates whether incorporating a PRS for CAD (PRS-CAD) into clinical decision-making improves cardiovascular risk stratification and leads to better primary prevention in individuals with intermediate estimated 10-year cardiovascular risk.

Participants aged 40-69 years with intermediate CVD risk based on the SCORE2 algorithm will be randomized 1:1 into two groups. In the intervention arm, the PRS-CAD will be calculated using a validated genome-wide algorithm and integrated with the SCORE2 risk to generate a combined PRS-CAD-SCORE2 estimate. Risk will be communicated to participants and their healthcare providers using a standardized, structured communication tool developed by the study team. Participants with elevated combined risk will be referred to lipid clinics for further evaluation. In the control arm, participants will receive standard SCORE2-based risk communication, without inclusion of genetic information.

All participants will receive written lifestyle guidance . Physicians will receive the results in a structured format.

The primary endpoint is the change in SCORE2 from baseline to 15 months. Secondary endpoints include changes in blood pressure, lipid levels, glucose, HbA1c, hs-CRP, BMI, weight, adherence to the Mediterranean diet (Predimed score), physical activity (IPAQ), tobacco abstinence, medication adherence (MARS), and psychological measures (DASS-21, motivation for change, satisfaction with risk communication). Prescription rates of statins and other preventive therapies, new diagnoses (e.g., diabetes), and new cardiovascular events will also be recorded. Epigenomic analyses will be conducted to explore interactions between genetic risk, lifestyle, and DNA methylation.

All outcomes will be assessed at 15 months with blinded outcome assessment. The study aims to inform the clinical utility of integrating PRS into preventive cardiovascular care and support the move toward personalized medicine in primary prevention.

ELIGIBILITY:
Inclusion Criteria:

* 40-69 years old
* Intermediate cardiovascular risk based on SCORE2 or SCORE2-Diabetes
* Able to give informed consent (understanding German or French or with an interpreter)
* Written Informed Consent

Exclusion Criteria:

* Patient treated under lipid-lowering therapy (defined as statin, ezetimib, bempedoïc acid, PCSK-9 inhibitors)
* History of previous cardiovascular disease: coronary artery disease (CAD), peripheral artery disease and ischemic stroke (including transitory ischemic stroke).
* Chronic kidney disease (CKD) define as an estimated glomerular filtration rate (eGFR) of less than 30 ml/min or less than 60 ml/min with albuminuria patients with diabetes and end organ damage (classified as very high risk according to ESC guidelines).
* Other participation in a clinical study related to CV risk or lifestyle interventions (e.g. diet, smoking cessation...)
* Life expectancy of less than one year

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in SCORE2 between baseline and 15 months | 15 months
  Mean change in SCORE2 cardiovascular risk score from baseline to 15-month follow-up, comparing the intervention (PRS-CAD + SCORE2) and control (SCORE2 only) arms.

SECONDARY OUTCOMES:
Change in systolic blood pressure | Baseline to 15 months
  Measured using validated automated oscillometric device at rest
Change in diastolic blood pressure | Baseline to 15 months
  Measured using validated automated oscillometric device at rest
Change in total cholesterol | Baseline to 15 months
  Measured via fasting venous blood sample
Change in HDL cholesterol (HDL-C) | Baseline to 15 months
  Measured via fasting venous blood sample
Change in LDL cholesterol (LDL-C) | Baseline to 15 months
  Measured via fasting venous blood sample
Change in triglyceride levels | Baseline to 15 months
  Measured via fasting venous blood sample
Change in fasting glucose | Baseline to 15 months
  Measured via fasting venous blood sample
Change in HbA1c | Baseline to 15 months
  Measured via venous blood sample
Change in high-sensitivity C-reactive protein (hs-CRP) | Baseline to 15 months
  Measured via fasting venous blood sample
Change in DNA methylation patterns | Baseline to 15 months
  Assessment of genome-wide DNA methylation changes from peripheral blood samples. DNA methylation will be analyzed in relation to adherence to the Mediterranean diet (measured via Predimed 14-item questionnaire) and its interaction with polygenic risk scores for coronary artery disease.
Tobacco abstinence status | Baseline to 15 months
  Self-reported smoking status assessed at follow-up
Change in body mass index (BMI) | Baseline to 15 months
  Calculated using measured weight and height (kg/m²)
Change in body weight | Baseline to 15 months
  Measured in kilograms using calibrated scale
Change in dietary adherence | Baseline to 15 months
  Measured by the Predimed 14-item questionnaire (score range: 0-14; higher scores indicate greater adherence to the Mediterranean diet)
Change in physical activity level | Baseline to 15 months
  Assessed using the International Physical Activity Questionnaire (IPAQ, long form; score expressed in MET-minutes/week; higher values indicate greater physical activity).
Change in medication adherence | Baseline to 15 months
  Assessed using the Medication Adherence Report Scale (MARS, 5-item version) score range: 5-25; higher scores indicate better adherence.
Change in motivation for lifestyle change | Baseline to 15 months
  Measured using the 32-item Readiness for Change Questionnaire; score range depends on subscale (e.g., Precontemplation, Contemplation, Action); higher scores indicate greater readiness for behavior change.
Change in psychological well-being | Baseline to 15 months
  Assessed using the Depression Anxiety Stress Scale (DASS-21); each subscale score ranges from 0 to 42, with higher scores indicating greater severity of symptoms.
Participant satisfaction with the intervention | Baseline to 15 months
  Measured via structured self-reported survey on a 5-point Likert scale (1 = not satisfied at all, 5 = very satisfied).
Number of visits to healthcare providers (HCPs) | Baseline to 15 months
  Self-reported and verified via medical records when available
Initiation of new statin therapy | Baseline to 15 months
  Number of participants with newly prescribed statins during follow-up period
Initiation of new antihypertensive therapy | Baseline to 15 months
  Number of participants with newly prescribed antihypertensive medications during follow-up period
Initiation of new antidiabetic therapy | Baseline to 15 months
  Number of participants with newly prescribed antidiabetic medications (oral or injectable) during follow-up period
Incidence of new cardiovascular events | Baseline to 15 months
  Number of participants with new cardiovascular events defined as new diagnosis of myocardial infarction, stroke, or other major adverse cardiovascular event (MACE); verified through clinical records
Incidence of newly diagnosed diabetes mellitus | Baseline to 15 months
  Number of participants with newly diagnosed type 2 diabetes confirmed by GP or medical record during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Rodondi, MD, Study Chair — University hospital of Bern
Locations (2):
- Switzerland (2):
  - University of Bern, Institute of Primary Health Care (BIHAM), Bern
  - University of Lausanne, Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared after official request

REFERENCES:
- [Background] De Montmollin M, Betrisey S, Feller M, Moutzouri E, Blum MR, Amsler J, Papazoglou DD, Moller B, Rodondi N. Achilles tendon ultrasonography in the clinical screening of familial hypercholesterolaemia - a cross-sectional analysis. Swiss Med Wkly. 2023 Nov 20;153:40127. doi: 10.57187/smw.2023.40127. PMID 37984334
- [Background] Ripatti P, Ramo JT, Mars NJ, Fu Y, Lin J, Soderlund S, Benner C, Surakka I, Kiiskinen T, Havulinna AS, Palta P, Freimer NB, Widen E, Salomaa V, Tukiainen T, Pirinen M, Palotie A, Taskinen MR, Ripatti S; FinnGendagger. Polygenic Hyperlipidemias and Coronary Artery Disease Risk. Circ Genom Precis Med. 2020 Apr;13(2):e002725. doi: 10.1161/CIRCGEN.119.002725. Epub 2020 Mar 10. PMID 32154731
- [Background] Jeemon P, Harikrishnan S, Sanjay G, Sivasubramonian S, Lekha TR, Padmanabhan S, Tandon N, Prabhakaran D. A PROgramme of Lifestyle Intervention in Families for Cardiovascular risk reduction (PROLIFIC Study): design and rationale of a family based randomized controlled trial in individuals with family history of premature coronary heart disease. BMC Public Health. 2017 Jan 5;17(1):10. doi: 10.1186/s12889-016-3928-6. PMID 28056897
- [Background] Lindbohm JV, Sipila PN, Mars N, Knuppel A, Pentti J, Nyberg ST, Frank P, Ahmadi-Abhari S, Brunner EJ, Shipley MJ, Singh-Manoux A, Tabak AG, Batty GD, Kivimaki M. Association between change in cardiovascular risk scores and future cardiovascular disease: analyses of data from the Whitehall II longitudinal, prospective cohort study. Lancet Digit Health. 2021 Jul;3(7):e434-e444. doi: 10.1016/S2589-7500(21)00079-0. PMID 34167764
- [Background] Willis A, Davies M, Yates T, Khunti K. Primary prevention of cardiovascular disease using validated risk scores: a systematic review. J R Soc Med. 2012 Aug;105(8):348-56. doi: 10.1258/jrsm.2012.110193. PMID 22907552
- [Background] Schwalm JD, McCready T, Lopez-Jaramillo P, Yusoff K, Attaran A, Lamelas P, Camacho PA, Majid F, Bangdiwala SI, Thabane L, Islam S, McKee M, Yusuf S. A community-based comprehensive intervention to reduce cardiovascular risk in hypertension (HOPE 4): a cluster-randomised controlled trial. Lancet. 2019 Oct 5;394(10205):1231-1242. doi: 10.1016/S0140-6736(19)31949-X. Epub 2019 Sep 2. PMID 31488369
- [Background] Daumit GL, Dalcin AT, Dickerson FB, Miller ER, Evins AE, Cather C, Jerome GJ, Young DR, Charleston JB, Gennusa JV 3rd, Goldsholl S, Cook C, Heller A, McGinty EE, Crum RM, Appel LJ, Wang NY. Effect of a Comprehensive Cardiovascular Risk Reduction Intervention in Persons With Serious Mental Illness: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e207247. doi: 10.1001/jamanetworkopen.2020.7247. PMID 32530472
- [Background] SCORE2 working group and ESC Cardiovascular risk collaboration. SCORE2 risk prediction algorithms: new models to estimate 10-year risk of cardiovascular disease in Europe. Eur Heart J. 2021 Jul 1;42(25):2439-2454. doi: 10.1093/eurheartj/ehab309. PMID 34120177
- [Background] Mohananey A, Tseng AS, Julakanti RR, Gonzalez-Bonilla HM, Kruisselbrink T, Prochnow C, Rodman S, Lin G, Redfield MM, Rosenbaum AN, Pereira NL. An intervention strategy to improve genetic testing for dilated cardiomyopathy in a heart failure clinic. Genet Med. 2023 Mar;25(3):100341. doi: 10.1016/j.gim.2022.11.009. Epub 2022 Dec 6. PMID 36472615
- [Background] Shefer G, Silarova B, Usher-Smith J, Griffin S. The response to receiving phenotypic and genetic coronary heart disease risk scores and lifestyle advice - a qualitative study. BMC Public Health. 2016 Dec 3;16(1):1221. doi: 10.1186/s12889-016-3867-2. PMID 27914472
- [Background] Brockman DG, Petronio L, Dron JS, Kwon BC, Vosburg T, Nip L, Tang A, O'Reilly M, Lennon N, Wong B, Ng K, Huang KH, Fahed AC, Khera AV. Design and user experience testing of a polygenic score report: a qualitative study of prospective users. BMC Med Genomics. 2021 Oct 1;14(1):238. doi: 10.1186/s12920-021-01056-0. PMID 34598685
- [Background] Viigimaa M, Jurisson M, Pisarev H, Kalda R, Alavere H, Irs A, Saar A, Fischer K, Lall K, Kruuv-Kao K, Mars N, Widen E, Ripatti S, Metspalu A. Effectiveness and feasibility of cardiovascular disease personalized prevention on high polygenic risk score subjects: a randomized controlled pilot study. Eur Heart J Open. 2022 Dec 15;2(6):oeac079. doi: 10.1093/ehjopen/oeac079. eCollection 2022 Nov. PMID 36600884
- [Background] Knowles JW, Zarafshar S, Pavlovic A, Goldstein BA, Tsai S, Li J, McConnell MV, Absher D, Ashley EA, Kiernan M, Ioannidis JPA, Assimes TL. Impact of a Genetic Risk Score for Coronary Artery Disease on Reducing Cardiovascular Risk: A Pilot Randomized Controlled Study. Front Cardiovasc Med. 2017 Aug 14;4:53. doi: 10.3389/fcvm.2017.00053. eCollection 2017. PMID 28856136
- [Background] Silarova B, Sharp S, Usher-Smith JA, Lucas J, Payne RA, Shefer G, Moore C, Girling C, Lawrence K, Tolkien Z, Walker M, Butterworth A, Di Angelantonio E, Danesh J, Griffin SJ. Effect of communicating phenotypic and genetic risk of coronary heart disease alongside web-based lifestyle advice: the INFORM Randomised Controlled Trial. Heart. 2019 Jul;105(13):982-989. doi: 10.1136/heartjnl-2018-314211. Epub 2019 Mar 30. PMID 30928969
- [Background] Kumuthini J, Zick B, Balasopoulou A, Chalikiopoulou C, Dandara C, El-Kamah G, Findley L, Katsila T, Li R, Maceda EB, Monye H, Rada G, Thong MK, Wanigasekera T, Kennel H, Marimuthu V; G2MC Evidence investigators; Williams MS, Al-Mulla F, Abramowicz M. The clinical utility of polygenic risk scores in genomic medicine practices: a systematic review. Hum Genet. 2022 Nov;141(11):1697-1704. doi: 10.1007/s00439-022-02452-x. Epub 2022 Apr 30. PMID 35488921
- [Background] King A, Wu L, Deng HW, Shen H, Wu C. Polygenic risk score improves the accuracy of a clinical risk score for coronary artery disease. BMC Med. 2022 Nov 7;20(1):385. doi: 10.1186/s12916-022-02583-y. PMID 36336692
- [Background] O'Sullivan JW, Raghavan S, Marquez-Luna C, Luzum JA, Damrauer SM, Ashley EA, O'Donnell CJ, Willer CJ, Natarajan P; American Heart Association Council on Genomic and Precision Medicine; Council on Clinical Cardiology; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Radiology and Intervention; Council on Lifestyle and Cardiometabolic Health; and Council on Peripheral Vascular Disease. Polygenic Risk Scores for Cardiovascular Disease: A Scientific Statement From the American Heart Association. Circulation. 2022 Aug 23;146(8):e93-e118. doi: 10.1161/CIR.0000000000001077. Epub 2022 Jul 18. PMID 35862132
- [Background] Sud A, Horton RH, Hingorani AD, Tzoulaki I, Turnbull C, Houlston RS, Lucassen A. Realistic expectations are key to realising the benefits of polygenic scores. BMJ. 2023 Feb 28;380:e073149. doi: 10.1136/bmj-2022-073149. PMID 36854461
- [Background] Klarin D, Natarajan P. Clinical utility of polygenic risk scores for coronary artery disease. Nat Rev Cardiol. 2022 May;19(5):291-301. doi: 10.1038/s41569-021-00638-w. Epub 2021 Nov 22. PMID 34811547
- [Background] Natarajan P, Young R, Stitziel NO, Padmanabhan S, Baber U, Mehran R, Sartori S, Fuster V, Reilly DF, Butterworth A, Rader DJ, Ford I, Sattar N, Kathiresan S. Polygenic Risk Score Identifies Subgroup With Higher Burden of Atherosclerosis and Greater Relative Benefit From Statin Therapy in the Primary Prevention Setting. Circulation. 2017 May 30;135(22):2091-2101. doi: 10.1161/CIRCULATIONAHA.116.024436. Epub 2017 Feb 21. PMID 28223407
- [Background] Mega JL, Stitziel NO, Smith JG, Chasman DI, Caulfield M, Devlin JJ, Nordio F, Hyde C, Cannon CP, Sacks F, Poulter N, Sever P, Ridker PM, Braunwald E, Melander O, Kathiresan S, Sabatine MS. Genetic risk, coronary heart disease events, and the clinical benefit of statin therapy: an analysis of primary and secondary prevention trials. Lancet. 2015 Jun 6;385(9984):2264-2271. doi: 10.1016/S0140-6736(14)61730-X. Epub 2015 Mar 4. PMID 25748612
- [Background] Mars N, Koskela JT, Ripatti P, Kiiskinen TTJ, Havulinna AS, Lindbohm JV, Ahola-Olli A, Kurki M, Karjalainen J, Palta P; FinnGen; Neale BM, Daly M, Salomaa V, Palotie A, Widen E, Ripatti S. Polygenic and clinical risk scores and their impact on age at onset and prediction of cardiometabolic diseases and common cancers. Nat Med. 2020 Apr;26(4):549-557. doi: 10.1038/s41591-020-0800-0. Epub 2020 Apr 7. PMID 32273609
- [Background] Aragam KG, Dobbyn A, Judy R, Chaffin M, Chaudhary K, Hindy G, Cagan A, Finneran P, Weng LC, Loos RJF, Nadkarni G, Cho JH, Kember RL, Baras A, Reid J, Overton J, Philippakis A, Ellinor PT, Weiss ST, Rader DJ, Lubitz SA, Smoller JW, Karlson EW, Khera AV, Kathiresan S, Do R, Damrauer SM, Natarajan P. Limitations of Contemporary Guidelines for Managing Patients at High Genetic Risk of Coronary Artery Disease. J Am Coll Cardiol. 2020 Jun 9;75(22):2769-2780. doi: 10.1016/j.jacc.2020.04.027. PMID 32498804
- [Background] Inouye M, Abraham G, Nelson CP, Wood AM, Sweeting MJ, Dudbridge F, Lai FY, Kaptoge S, Brozynska M, Wang T, Ye S, Webb TR, Rutter MK, Tzoulaki I, Patel RS, Loos RJF, Keavney B, Hemingway H, Thompson J, Watkins H, Deloukas P, Di Angelantonio E, Butterworth AS, Danesh J, Samani NJ; UK Biobank CardioMetabolic Consortium CHD Working Group. Genomic Risk Prediction of Coronary Artery Disease in 480,000 Adults: Implications for Primary Prevention. J Am Coll Cardiol. 2018 Oct 16;72(16):1883-1893. doi: 10.1016/j.jacc.2018.07.079. PMID 30309464
- [Background] Musliner KL, Mortensen PB, McGrath JJ, Suppli NP, Hougaard DM, Bybjerg-Grauholm J, Baekvad-Hansen M, Andreassen O, Pedersen CB, Pedersen MG, Mors O, Nordentoft M, Borglum AD, Werge T, Agerbo E; Bipolar Disorder Working Group of the Psychiatric Genomics Consortium. Association of Polygenic Liabilities for Major Depression, Bipolar Disorder, and Schizophrenia With Risk for Depression in the Danish Population. JAMA Psychiatry. 2019 May 1;76(5):516-525. doi: 10.1001/jamapsychiatry.2018.4166. PMID 30698613
- [Background] Muranen TA, Mavaddat N, Khan S, Fagerholm R, Pelttari L, Lee A, Aittomaki K, Blomqvist C, Easton DF, Nevanlinna H. Polygenic risk score is associated with increased disease risk in 52 Finnish breast cancer families. Breast Cancer Res Treat. 2016 Aug;158(3):463-9. doi: 10.1007/s10549-016-3897-6. Epub 2016 Jul 20. PMID 27438779
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Jun 18;139(25):e1046-e1081. doi: 10.1161/CIR.0000000000000624. Epub 2018 Nov 10. No abstract available. PMID 30565953
- [Background] Sposito AC, Ramires JA, Jukema JW, Molina JC, da Silva PM, Ghadanfar MM, Wilson PW. Physicians' attitudes and adherence to use of risk scores for primary prevention of cardiovascular disease: cross-sectional survey in three world regions. Curr Med Res Opin. 2009 May;25(5):1171-8. doi: 10.1185/03007990902846423. PMID 19323611
- [Background] Finnikin S, Ryan R, Marshall T. Statin initiations and QRISK2 scoring in UK general practice: a THIN database study. Br J Gen Pract. 2017 Dec;67(665):e881-e887. doi: 10.3399/bjgp17X693485. Epub 2017 Oct 23. PMID 29061715
- [Background] Delabays B, Marques-Vidal P, Kronenberg F, Waeber G, Vollenweider P, Vaucher J. Use of lipoprotein(a) for refining cardiovascular risk prediction in a low-risk population: The CoLaus/PsyCoLaus study. Eur J Prev Cardiol. 2021 Jul 23;28(8):e18-e20. doi: 10.1177/2047487320938271. Epub 2020 Jul 5. No abstract available. PMID 34298560
- [Background] Mosca L, Banka CL, Benjamin EJ, Berra K, Bushnell C, Dolor RJ, Ganiats TG, Gomes AS, Gornik HL, Gracia C, Gulati M, Haan CK, Judelson DR, Keenan N, Kelepouris E, Michos ED, Newby LK, Oparil S, Ouyang P, Oz MC, Petitti D, Pinn VW, Redberg RF, Scott R, Sherif K, Smith SC Jr, Sopko G, Steinhorn RH, Stone NJ, Taubert KA, Todd BA, Urbina E, Wenger NK; Expert Panel/Writing Group; American Heart Association; American Academy of Family Physicians; American College of Obstetricians and Gynecologists; American College of Cardiology Foundation; Society of Thoracic Surgeons; American Medical Women's Association; Centers for Disease Control and Prevention; Office of Research on Women's Health; Association of Black Cardiologists; American College of Physicians; World Heart Federation; National Heart, Lung, and Blood Institute; American College of Nurse Practitioners. Evidence-based guidelines for cardiovascular disease prevention in women: 2007 update. Circulation. 2007 Mar 20;115(11):1481-501. doi: 10.1161/CIRCULATIONAHA.107.181546. Epub 2007 Feb 19. No abstract available. PMID 17309915
- [Background] Edwards FH, Ferraris VA, Shahian DM, Peterson E, Furnary AP, Haan CK, Bridges CR; Society of Thoracic Surgeons. Gender-specific practice guidelines for coronary artery bypass surgery: perioperative management. Ann Thorac Surg. 2005 Jun;79(6):2189-94. doi: 10.1016/j.athoracsur.2005.02.065. PMID 15919346
- [Background] Maas AH, Appelman YE. Gender differences in coronary heart disease. Neth Heart J. 2010 Dec;18(12):598-602. doi: 10.1007/s12471-010-0841-y. PMID 21301622
- [Background] Damask A, Steg PG, Schwartz GG, Szarek M, Hagstrom E, Badimon L, Chapman MJ, Boileau C, Tsimikas S, Ginsberg HN, Banerjee P, Manvelian G, Pordy R, Hess S, Overton JD, Lotta LA, Yancopoulos GD, Abecasis GR, Baras A, Paulding C; Regeneron Genetics Center and the ODYSSEY OUTCOMES Investigators. Patients With High Genome-Wide Polygenic Risk Scores for Coronary Artery Disease May Receive Greater Clinical Benefit From Alirocumab Treatment in the ODYSSEY OUTCOMES Trial. Circulation. 2020 Feb 25;141(8):624-636. doi: 10.1161/CIRCULATIONAHA.119.044434. Epub 2019 Nov 11. PMID 31707832
- [Background] Marston NA, Kamanu FK, Nordio F, Gurmu Y, Roselli C, Sever PS, Pedersen TR, Keech AC, Wang H, Lira Pineda A, Giugliano RP, Lubitz SA, Ellinor PT, Sabatine MS, Ruff CT. Predicting Benefit From Evolocumab Therapy in Patients With Atherosclerotic Disease Using a Genetic Risk Score: Results From the FOURIER Trial. Circulation. 2020 Feb 25;141(8):616-623. doi: 10.1161/CIRCULATIONAHA.119.043805. Epub 2019 Nov 11. PMID 31707849
- [Background] Kullo IJ, Jouni H, Austin EE, Brown SA, Kruisselbrink TM, Isseh IN, Haddad RA, Marroush TS, Shameer K, Olson JE, Broeckel U, Green RC, Schaid DJ, Montori VM, Bailey KR. Incorporating a Genetic Risk Score Into Coronary Heart Disease Risk Estimates: Effect on Low-Density Lipoprotein Cholesterol Levels (the MI-GENES Clinical Trial). Circulation. 2016 Mar 22;133(12):1181-8. doi: 10.1161/CIRCULATIONAHA.115.020109. Epub 2016 Feb 25. PMID 26915630
- [Background] de La Harpe R, Thorball CW, Redin C, Fournier S, Muller O, Strambo D, Michel P, Vollenweider P, Marques-Vidal P, Fellay J, Vaucher J. Combining European and U.S. risk prediction models with polygenic risk scores to refine cardiovascular prevention: the CoLaus|PsyCoLaus Study. Eur J Prev Cardiol. 2023 May 9;30(7):561-571. doi: 10.1093/eurjpc/zwad012. PMID 36652418
- [Background] Elliott J, Bodinier B, Bond TA, Chadeau-Hyam M, Evangelou E, Moons KGM, Dehghan A, Muller DC, Elliott P, Tzoulaki I. Predictive Accuracy of a Polygenic Risk Score-Enhanced Prediction Model vs a Clinical Risk Score for Coronary Artery Disease. JAMA. 2020 Feb 18;323(7):636-645. doi: 10.1001/jama.2019.22241. PMID 32068818
- [Background] Sun L, Pennells L, Kaptoge S, Nelson CP, Ritchie SC, Abraham G, Arnold M, Bell S, Bolton T, Burgess S, Dudbridge F, Guo Q, Sofianopoulou E, Stevens D, Thompson JR, Butterworth AS, Wood A, Danesh J, Samani NJ, Inouye M, Di Angelantonio E. Polygenic risk scores in cardiovascular risk prediction: A cohort study and modelling analyses. PLoS Med. 2021 Jan 14;18(1):e1003498. doi: 10.1371/journal.pmed.1003498. eCollection 2021 Jan. PMID 33444330
- [Background] Khera AV, Chaffin M, Aragam KG, Haas ME, Roselli C, Choi SH, Natarajan P, Lander ES, Lubitz SA, Ellinor PT, Kathiresan S. Genome-wide polygenic scores for common diseases identify individuals with risk equivalent to monogenic mutations. Nat Genet. 2018 Sep;50(9):1219-1224. doi: 10.1038/s41588-018-0183-z. Epub 2018 Aug 13. PMID 30104762
- [Background] Khera AV, Emdin CA, Drake I, Natarajan P, Bick AG, Cook NR, Chasman DI, Baber U, Mehran R, Rader DJ, Fuster V, Boerwinkle E, Melander O, Orho-Melander M, Ridker PM, Kathiresan S. Genetic Risk, Adherence to a Healthy Lifestyle, and Coronary Disease. N Engl J Med. 2016 Dec 15;375(24):2349-2358. doi: 10.1056/NEJMoa1605086. Epub 2016 Nov 13. PMID 27959714
- [Background] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM, Binno S; ESC Scientific Document Group. 2016 European Guidelines on cardiovascular disease prevention in clinical practice: The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts)Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation (EACPR). Eur Heart J. 2016 Aug 1;37(29):2315-2381. doi: 10.1093/eurheartj/ehw106. Epub 2016 May 23. No abstract available. PMID 27222591
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC National Cardiac Societies; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur Heart J. 2021 Sep 7;42(34):3227-3337. doi: 10.1093/eurheartj/ehab484. No abstract available. PMID 34458905
- [Background] Mach F, Baigent C, Catapano AL, Koskinas KC, Casula M, Badimon L, Chapman MJ, De Backer GG, Delgado V, Ference BA, Graham IM, Halliday A, Landmesser U, Mihaylova B, Pedersen TR, Riccardi G, Richter DJ, Sabatine MS, Taskinen MR, Tokgozoglu L, Wiklund O; ESC Scientific Document Group. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. Eur Heart J. 2020 Jan 1;41(1):111-188. doi: 10.1093/eurheartj/ehz455. No abstract available. PMID 31504418
- [Background] Silverman MG, Ference BA, Im K, Wiviott SD, Giugliano RP, Grundy SM, Braunwald E, Sabatine MS. Association Between Lowering LDL-C and Cardiovascular Risk Reduction Among Different Therapeutic Interventions: A Systematic Review and Meta-analysis. JAMA. 2016 Sep 27;316(12):1289-97. doi: 10.1001/jama.2016.13985. PMID 27673306
- [Background] Lozano R, Naghavi M, Foreman K, Lim S, Shibuya K, Aboyans V, Abraham J, Adair T, Aggarwal R, Ahn SY, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Barker-Collo S, Bartels DH, Bell ML, Benjamin EJ, Bennett D, Bhalla K, Bikbov B, Bin Abdulhak A, Birbeck G, Blyth F, Bolliger I, Boufous S, Bucello C, Burch M, Burney P, Carapetis J, Chen H, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahodwala N, De Leo D, Degenhardt L, Delossantos A, Denenberg J, Des Jarlais DC, Dharmaratne SD, Dorsey ER, Driscoll T, Duber H, Ebel B, Erwin PJ, Espindola P, Ezzati M, Feigin V, Flaxman AD, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabriel SE, Gakidou E, Gaspari F, Gillum RF, Gonzalez-Medina D, Halasa YA, Haring D, Harrison JE, Havmoeller R, Hay RJ, Hoen B, Hotez PJ, Hoy D, Jacobsen KH, James SL, Jasrasaria R, Jayaraman S, Johns N, Karthikeyan G, Kassebaum N, Keren A, Khoo JP, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lipnick M, Lipshultz SE, Ohno SL, Mabweijano J, MacIntyre MF, Mallinger L, March L, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGrath J, Mensah GA, Merriman TR, Michaud C, Miller M, Miller TR, Mock C, Mocumbi AO, Mokdad AA, Moran A, Mulholland K, Nair MN, Naldi L, Narayan KM, Nasseri K, Norman P, O'Donnell M, Omer SB, Ortblad K, Osborne R, Ozgediz D, Pahari B, Pandian JD, Rivero AP, Padilla RP, Perez-Ruiz F, Perico N, Phillips D, Pierce K, Pope CA 3rd, Porrini E, Pourmalek F, Raju M, Ranganathan D, Rehm JT, Rein DB, Remuzzi G, Rivara FP, Roberts T, De Leon FR, Rosenfeld LC, Rushton L, Sacco RL, Salomon JA, Sampson U, Sanman E, Schwebel DC, Segui-Gomez M, Shepard DS, Singh D, Singleton J, Sliwa K, Smith E, Steer A, Taylor JA, Thomas B, Tleyjeh IM, Towbin JA, Truelsen T, Undurraga EA, Venketasubramanian N, Vijayakumar L, Vos T, Wagner GR, Wang M, Wang W, Watt K, Weinstock MA, Weintraub R, Wilkinson JD, Woolf AD, Wulf S, Yeh PH, Yip P, Zabetian A, Zheng ZJ, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Global and regional mortality from 235 causes of death for 20 age groups in 1990 and 2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2095-128. doi: 10.1016/S0140-6736(12)61728-0. PMID 23245604
- [Background] Wang F, Yu Y, Mubarik S, Zhang Y, Liu X, Cheng Y, Yu C, Cao J. Global Burden of Ischemic Heart Disease and Attributable Risk Factors, 1990-2017: A Secondary Analysis Based on the Global Burden of Disease Study 2017. Clin Epidemiol. 2021 Sep 21;13:859-870. doi: 10.2147/CLEP.S317787. eCollection 2021. PMID 34584461
- See also: UK government consultation paper outlining a national strategy to shift healthcare towards prevention, including the potential role of genomics and polygenic risk scores in personalized disease prevention. — https://www.gov.uk/government/consultations/advancing-our-health-prevention-in-the-2020s/advancing-our-health-prevention-in-the-2020s-consultation-document
- See also: Heart Age Calculator — https://www.heartfoundation.org.au/heart-age-calculator
- See also: Readiness for Change Questionnaire — http://tmctohealth.com/wp-content/uploads/2017/03/TMC-To-Health_Readiness-for-Change-Questionnaire.pdf.